CLINICAL TRIAL: NCT04579861
Title: Determining Post-operative Morbidity and Mortality Following Gynaecological Oncology Surgery: a Multicentre, International, Prospective Cohort Study Led by the Global Gynaecological Oncology Surgical Outcomes Collaborative (GO SOAR)
Brief Title: GO SOAR1: Post-Operative Morbidity and Mortality Following Gynaecological Oncology Surgery
Acronym: GO SOAR1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Faiza Gaba (Other Government)
Collaborators: University of Aberdeen (Other); University of Hertfordshire (Other); NHS Grampian (Other Government); Queen Mary University of London (Other); European Network of Young Gynae Oncologists (Unknown); Society of Gynecologic Oncology (Other); Cancer Diseases Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Faiza Gaba, Collaborative Lead & Chief Investigator, NHS Grampian
Organization: NHS Grampian (Other Government)
Other Study IDs: 5009
Record Dates: First submitted 2020-09-29; First posted 2020-10-08 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Gynecologic Cancer; Surgery; Surgery--Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High human development: Countries classified as very high and high human development as per the United Nations development programme.
  Interventions: Other: Prospective data collection following gynaecological oncology surgery
- Low and medium human development: Countries classified as low and medium human development as per the United Nations development programme.
  Interventions: Other: Prospective data collection following gynaecological oncology surgery

INTERVENTIONS:
Other: Prospective data collection following gynaecological oncology surgery — Prospective data collection and entry on database following gynaecological oncology surgery

SUMMARY:
The Global Gynaecological Oncology Surgical Outcomes Collaborative (GO SOAR) will develop a network of gynaecological oncology surgeons, surgical departments and other interested parties that will have the long-term ability to collaborate on outcome studies. The aims of the Collaborative are to:

1. Set the research agenda through research prioritisation in gynaecological oncology surgical outcomes.
2. Gather high quality data via a centralised database accessible to all sites that perform gynaecological oncology surgery.
3. Build sustainable international research by producing protocols/guidelines.
4. Train the researchers and leaders of tomorrow by providing open access to all GO SOAR training materials.

The Collaborative will lead to several studies.

The first GO SOAR collaborative study (GO SOAR1) will evaluate international variation of post-operative morbidity and mortality following gynaecological oncology surgery between country groups defined by the human development index (HDI).

DETAILED DESCRIPTION:
Study hypothesis

There is no variation in post-operative morbidity and mortality rates following gynaecological oncology surgery between HDI country groups.

Regulatory approval

Quality Improvement & Assurance Team, Research and Development NHS Grampian (Project ID 5009).

Study design

International, multi-centre, prospective cohort study.

Primary objectives

1. To evaluate international variation of post-operative morbidity and mortality following gynaecological oncology surgery between country groups defined by HDI.

Secondary objectives

1. To evaluate international variation between HDI country groups of intra-operative morbidity and mortality following gynaecological oncology surgery.
2. To evaluate international variation between HDI country groups of histological clearance rates of gynaecological malignancies.
3. To establish an international gynaecological oncology collaborative and surgical outcomes database.
4. To identify modifiable surgical processes.
5. To establish best practices and standards for gynaecological oncology surgery.
6. To champion promotion of quality improvement and research and gynaecological oncology surgical training.

Interventions

Patient data will be collected over a consecutive thirty day period through gynaecological oncology multidisciplinary teams/tumour boards and clinics across different human development index country groups. Additional data entry (beyond thirty days) is encouraged and may take place at the discretion of the participating site. All patients are followed up as per local protocols for thirty days post-operatively to identify post-surgical morbidity/mortality. For each patient, data will be captured on demographic variables, centre/unit/hospital site, FIGO staging, surgical modality, intra-operative morbidity/mortality, 30 day morbidity/mortality following surgery, tumour resectability, access to diagnostic endoscopy/hysteroscopy, histopathology/radiological imaging/laboratories/critical care facilities, multidisciplinary team/tumour board meetings, chemotherapy, radiotherapy seniority and training of lead surgeon. All data is collected on a customised, secure, password protected central REDCap database.

Follow up

All investigators are required to monitor patients for thirty days post-operatively to identify complications. Most of these events are expected to occur during the individual's inpatient stay. Centres must be proactive in identifying post-operative events (or an absence of them), within the limits of normal follow up. Local arrangements may include:

1. Daily review of patient status and notes before discharge to identify inpatient complications.
2. Reviewing the patient status at a post-surgery follow up appointment in an outpatient clinic or via telephone (if this is normal practice).
3. Checking hospital records (electronic/paper) or handover lists for re-attendances/re-admissions.
4. Checking for Emergency Department re-attendances.
5. Contacting general/family practitioners to enquire about complications managed in primary care.

International Steering Committee

An international steering committee will oversee the study. The committee will monitor and supervise progress and adherence to protocol. The committee will review at regular intervals relevant information from other sources, e.g. other audits/studies. It will ensure that the study is conducted to a high standard in line with Guidelines for Good Clinical Practice. The committee will meet every six months though more frequent meetings may be called if necessary. Meetings will be called for by the chief investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged >18 years undergoing curative, curative attempted but then abandoned (i.e. open/close laparotomy) or palliative surgery for primary tubo-ovarian/peritoneal, endometrial, cervical, vulval, vaginal, gestational trophoblastic malignancies.
2. Surgery for recurrent primary tubo-ovarian/peritoneal, endometrial, cervical, vulval, vaginal, gestational trophoblastic malignancies.
3. Open, minimal access (laparoscopic/robotic), minimal access converted to open or vaginal surgeries for tubo-ovarian/peritoneal, endometrial, cervical, vulval, vagina, gestational trophoblastic malignancies.
4. Elective and emergency surgeries.
5. Surgeries where pre-operative pathology thought to be benign but malignancy confirmed on histopathology post-operatively.

Exclusion Criteria:

1. Surgeries where pre-operative pathology thought to be malignant but benign disease confirmed on histopathology post-operatively.
2. Non gynaecological disease as the primary malignancy.
3. Diagnostic procedures (e.g. staging laparoscopy, image guided biopsy).
4. Any procedure not requiring a skin incision under general/regional anaesthesia (e.g. chemotherapy, radiotherapy, hysteroscopy).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women >18 years undergoing gynaecological oncology surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2021-01-19 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-operative surgical morbidity | 30 days
  Post-operative surgical morbidity
Post-operative surgical mortality | 30 days
  Post-operative surgical mortality

CONTACTS AND LOCATIONS:
Overall Officials: Faiza Gaba, Principal Investigator — NHS Grampian
Locations (1):
- NHS Grampian, Aberdeen, County (optional), United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaba F, Bizzarri N, Kamfwa P, Saiz A, Blyuss O, Paranjothy S, Ramirez PT, Cibula D; GO SOAR Team. Determining post-operative morbidity and mortality following gynecological oncology surgery: protocol for a multicenter, international, prospective cohort study (Global Gynaecological Oncology Surgical Outcomes Collaborative-GO SOAR). Int J Gynecol Cancer. 2021 Sep;31(9):1287-1291. doi: 10.1136/ijgc-2021-002586. PMID 34489356